CLINICAL TRIAL: NCT01659437
Title: Randomized Controlled Trial Comparing Efficacy of 8 Weeks Treatment With Clarithromycin and Rifampicin Versus Streptomycin and Rifampicin for Buruli Ulcer (M. Ulcerans Infection)
Brief Title: WHO Drug Study for Buruli Ulcer - Comparison of SR8 and CR8
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: University of Groningen (Other); Faculté de Médecine P&M Curie, Paris-6 - Site Pitié-Salpêtrière, France (Unknown); Drugs for Neglected Diseases (Other); World Alliance for Wound and Lymphoedema Care, Switzerland (Unknown); Inserm U892/CNRS 699 bactériologie, Université CHU;Angers- IRIS France (Unknown); Institute of Tropical Medicine, Antwerp, Belgium (Unknown); National Buruli ulcer Control Programme, Ghana Health Service, Accra, Ghana (Unknown); School of Med Sciences, Kwame Nkrumah Univ of Sci & Techn, Kumasi, Ghana (Unknown); Komfo Anokye Teaching Hospital (Other); Kumasi Center for Collaborative Research into Tropical Medicine, Kumasi, Ghana (Unknown); Plastic Surgery and Burns Centre, Korle-Bu Teaching Hospital, Accra, Ghana (Unknown); University of Ghana (Other); Noguchi Memorial Institute of Medical Research, Accra, Ghana (Unknown); Program Nat de Lutte contre la Lèpre et l'UB;Ulcère de Buruli, Cotonou, Benin (Unknown)
Responsible Party: Principal Investigator, Tjip van der Werf, Professor, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: T9-370-1
Record Dates: First submitted 2012-08-02; First posted 2012-08-07 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Mycobacterium Ulcerans Infection
Keywords: M. ulcerans; Buruli ulcer; drug trial; clarithromycin
MeSH Terms: conditions — Buruli Ulcer

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SR8 (Active Comparator): Streptomycin (S: 15 mg/kg per day, intramuscularly) in combination with rifampicin (R: 10 mg/kg per day, orally) for 8 weeks
  Interventions: Drug: Streptomycin intramuscular injection
- CR8 (Experimental): Clarithromycin (C: 15 mg/kg per day, oral extended release formulation) in combination with rifampicin (10 mg/kg per day, orally) for 8 weeks
  Interventions: Drug: Clarithromycin Extended Release

INTERVENTIONS:
Drug: Clarithromycin Extended Release — oral administration of Clarithromycin extended release
  Arms: CR8
Drug: Streptomycin intramuscular injection — daily intramuscular drug injection
  Arms: SR8

SUMMARY:
This is a WHO-sponsored trial.

Combination therapy with streptomycin and rifampicin has been the standard antibiotic treatment for M. ulcerans infection since 2004. In March 2010, a WHO Technical Advisory Group recommended that a trial be carried out to develop a fully oral treatment for the disease. Although the current treatment is effective, injection with streptomycin is a problem. Several small observational studies (published and unpublished) have shown that a fully oral treatment is promising.

This WHO sponsored study will be a randomized, controlled open label non-inferiority phase II/III, multi-centre trial (1 centre in Benin and 4 centres in Ghana), with two parallel treatment groups. The ultimate goal is to search for an effective alternative treatment to the current standard WHO-recommended therapy for all forms of Buruli ulcer, which includes injections of streptomycin with inherent logistic, operational and safety disadvantages.

Financial and material support:

1. American Leprosy Missions, USA
2. Raoul Follereau Foundation, France
3. MAP International, USA
4. Sanofi, France
5. 7th Framework Programme of the European Union: BuruliVac project (241500)
6. Aranz Medical Limited, New Zealand

DETAILED DESCRIPTION:
A total of 415 patients in whom Buruli ulcer has been clinically diagnosed will be included in the study, which will consist of 332 cases of category I and II Buruli ulcers (<10 cm) confirmed by polymerase chain reaction (PCR), plus 83 non PCR-confirmed Buruli ulcers. Patients will be randomized to receive treatment with the two antibiotic regimens as follows:

(i) Regimen I (SR8): 15 mg/kg streptomycin per day intramuscular injection for 8 weeks plus 10 mg/kg per day oral rifampicin for 8 weeks; (ii) Regimen II (CR8): 15 mg/kg per day oral extended-release clarithromycin for 8 weeks plus 10 mg/kg per day oral rifampicin for 8 weeks.

Assessments before, during and after the course of antibiotic treatment will include full medical history, clinical assessments and monitoring of vital signs, assessment of the lesion, laboratory investigations, hearing test, electrocardiogram, pregnancy test, voluntary HIV counseling and testing, and functional limitation assessment. The primary efficacy parameters are healing without recurrence and without excision surgery 12 months after the start of treatment.

The primary endpoint will be assessed by a panel of experts unaware of the treatment ('single blinded' for treatment allocation).

Statistician:

Mr Bruno Scherrer, Consultant, Drugs for Neglected Diseases initiative, Switzerland

Data Management:

Mr Raymond Omollo, Drugs for Neglected Diseases initiative (DNDi) Africa

ELIGIBILITY:
Inclusion criteria:

* All patients (both genders) with a clinical diagnosis of BUD (categories: I and II, cross-sectional diameter ≤ 10cm) as agreed by study site treatment team led by the lead clinicians

Exclusion criteria:

1. Patients with lesion sizes >10cm in cross-sectional diameter
2. Children < 5 years, or < 20 kilograms body weight
3. Pregnancy (self-reported, clinically diagnosed, or urine test (beta-hCG) positive
4. Patients with previous treatment of Buruli ulcer, tuberculosis or leprosy with at least one of the study drugs (rifampicin, streptomycin, clarithromycin)
5. Patients with history of hypersensitivity to rifampicin and/or streptomycin and/or clarithromycin
6. Patients with previous treatment with macrolide or quinolone antibiotics, or antituberculosis medication, or immuno-modulatory drugs including corticosteroids within one month
7. Patients with current treatment with any drugs likely to interact with the study medication, e.g, anticoagulants, cyclosporin, phenytoin, and phenobarbitone. Users of oral contraceptives should be notified that such contraceptive is less reliable if taken with rifampicin; alternative (mechanical) contraceptive methods will be discussed with the study participant
8. Patients with co-infection with HIV
9. Patients with history or having current clinical signs of ascites, jaundice, partial or complete deafness, myasthenia gravis, renal dysfunction (known or suspected), diabetes mellitus, and severe immune compromise (e.g., immunosuppressive drugs after organ transplant), or evidence of (previous) tuberculosis, Buruli ulcer or leprosy; or terminal illness (e.g., metastasized cancer)
10. Patients who are unable to take oral medication or having gastrointestinal disease likely to interfere with drug absorption
11. Patients with known or suspected bowel strictures who cannot tolerate macrolide antibiotics such as clarithromycin
12. Patients with mental condition, including addiction with substance abuse (alcohol, qat, etc) likely to interfere with possibility to comply with the study protocol
13. Patients who are not willing to give informed pre-consent, and consent (patient and/or parent/legal representative), or withdrawal of consent

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2012-12; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
healing without recurrence and without excision surgery | 12 months after start of treatment
  complete epithelialisation and absence of swelling at the site of original infection, measured 12 months after start of treatment; lesion site will be examined by inspection and palpation, and documented by digital camera; digital images will be examined by panel of wound experts unaware of treatment allocation

SECONDARY OUTCOMES:
Recurrence rate within 12 months of treatment initiation | 12 months
  number of recurrent lesions occurring after initial healing within 12 months after start of treatment
Rate of treatment failure within 12 months of treatment initiation | 12 months
  proportion of treatment failure will be compared between groups
Rate of paradoxical response within 12 months of treatment initiation | 12 months
  paradoxical responses that have occurred during BUD treatment will be compared in both treatment arms
Proportion of patients with reduction in lesion surface area within 12 months of treatment initiation | 12 months
  if not cured, will there be a difference between groups in terms of reduction of lesion size?
Time taken for complete lesion healing within 12 months of treatment initiation | 12 months
  do lesions heal faster in one of the two treatments?
Proportion (%) of patients with complete healing without additional surgery or relapse | 12 months
Interval between healing and recurrence | 12 months
  if recurrences occur, there might be a difference in time between healing and recurrences between treatment groups
Proportion of each type of surgery within 12 months of treatment initiation | 12 months
  We do not expect surgery but IF doctors operate, which type of surgery would doctors use, and does this differ between groups?
Time from treatment initiation to surgery if any | 12months
  does the timing of surgery differ between groups for the proportion of patients in whom doctors decide to operate?
Proportion of patients with residual functional limitations | 12 months
  do treatments differ in terms of chance to develop functional limitations?
Treatment discontinuation and compliance rates | 8 weeks
  one treatment might be better tolerated than the other; do treatments differ in terms of adherence problems, and do participants in any of these two treatment arms differ in terms of the chance to discontinue the treatment?
Incidence of all adverse effects (AEs) within 12 months of treatment initiation | 12 months
  adverse effects occurring during or after treatment may be different between treatments

CONTACTS AND LOCATIONS:
Overall Officials: Tjip S van der Werf, MD, PhD, Principal Investigator — University of Groningen, University Medical Centre Groningen; Richard O Phillips, MD, PhD, Study Director — Komfo Anokye Teaching Hospital, Kwame Nkrumah University of Science & Technology, Kumasi, Ghana; Annick Chauty, MD, Study Director — Pobè Health Centre, Pobè, Bénin; Kingsley B Asiedu, MD, MPH, Study Chair — WHO, GBUI, Geneva, Switserland
Locations (5):
- Pobè Treatment Center, Pobè, Benin
- Ghana (4):
  - Agogo Presbyterian Hospital, Agogo
  - Dunkwa Government Hospital, Dunkwa-on-Offin
  - Nkawie-Toase Government Hospital, Nkawie Panyin
  - Tepa Government Hosital, Tepa

IPD SHARING:
Plan to Share IPD: Yes
after publication, IPD will be made available at the time of publication; enrollment is complewted with 310 participants enrolled by Dec 2017; final report submitted for publication Sept 2019
Supporting Information: Study Protocol, SAP, ICF
Time Frame: data analysis report as well as data in OpenClinica deposited with DNDi Regional Africa Office Nairobi

REFERENCES:
- [Background] Nienhuis WA, Stienstra Y, Thompson WA, Awuah PC, Abass KM, Tuah W, Awua-Boateng NY, Ampadu EO, Siegmund V, Schouten JP, Adjei O, Bretzel G, van der Werf TS. Antimicrobial treatment for early, limited Mycobacterium ulcerans infection: a randomised controlled trial. Lancet. 2010 Feb 20;375(9715):664-72. doi: 10.1016/S0140-6736(09)61962-0. Epub 2010 Feb 3. PMID 20137805
- [Background] Chauty A, Ardant MF, Marsollier L, Pluschke G, Landier J, Adeye A, Goundote A, Cottin J, Ladikpo T, Ruf T, Ji B. Oral treatment for Mycobacterium ulcerans infection: results from a pilot study in Benin. Clin Infect Dis. 2011 Jan 1;52(1):94-6. doi: 10.1093/cid/ciq072. PMID 21148526
- [Background] Gordon CL, Buntine JA, Hayman JA, Lavender CJ, Fyfe JA, Hosking P, Starr M, Johnson PD. All-oral antibiotic treatment for buruli ulcer: a report of four patients. PLoS Negl Trop Dis. 2010 Nov 30;4(11):e770. doi: 10.1371/journal.pntd.0000770. No abstract available. PMID 21152060
- [Background] O'Brien DP, McDonald A, Callan P, Robson M, Friedman ND, Hughes A, Holten I, Walton A, Athan E. Successful outcomes with oral fluoroquinolones combined with rifampicin in the treatment of Mycobacterium ulcerans: an observational cohort study. PLoS Negl Trop Dis. 2012 Jan;6(1):e1473. doi: 10.1371/journal.pntd.0001473. Epub 2012 Jan 17. PMID 22272368
- [Derived] Phillips RO, Robert J, Abass KM, Thompson W, Sarfo FS, Wilson T, Sarpong G, Gateau T, Chauty A, Omollo R, Ochieng Otieno M, Egondi TW, Ampadu EO, Agossadou D, Marion E, Ganlonon L, Wansbrough-Jones M, Grosset J, Macdonald JM, Treadwell T, Saunderson P, Paintsil A, Lehman L, Frimpong M, Sarpong NF, Saizonou R, Tiendrebeogo A, Ohene SA, Stienstra Y, Asiedu KB, van der Werf TS; study team. Rifampicin and clarithromycin (extended release) versus rifampicin and streptomycin for limited Buruli ulcer lesions: a randomised, open-label, non-inferiority phase 3 trial. Lancet. 2020 Apr 18;395(10232):1259-1267. doi: 10.1016/S0140-6736(20)30047-7. Epub 2020 Mar 12. PMID 32171422
- [Derived] Converse PJ, Almeida DV, Tasneen R, Saini V, Tyagi S, Ammerman NC, Li SY, Anders NM, Rudek MA, Grosset JH, Nuermberger EL. Shorter-course treatment for Mycobacterium ulcerans disease with high-dose rifamycins and clofazimine in a mouse model of Buruli ulcer. PLoS Negl Trop Dis. 2018 Aug 13;12(8):e0006728. doi: 10.1371/journal.pntd.0006728. eCollection 2018 Aug. PMID 30102705
- See also: WHO Buruli ulcer website — http://www.who.int/buruli/en/